CLINICAL TRIAL: NCT04936867
Title: The CArdiac Imaging RegistrY Study: Computed ToMogrAphy for Risk Stratification and Diagnostic Safety
Brief Title: The CArdiac Imaging RegistrY Study
Acronym: CARYSMA
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Valentina Puentmann, Clinical professor, Johann Wolfgang Goethe University Hospital
Other Study IDs: CARYSMA Registry Study 466/16
Record Dates: First submitted 2021-06-16; First posted 2021-06-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective longitudinal observational investigator-led single centre cohort study we will include patients undergoing cardio-CT for clinical reasons, to evaluate the role of cardio-CT terms of its diagnostic and prognostic value, as well as risk-benefit ratio.

Particular aims include:

1. To determine the prevalence of CAD for age, gender, ethnicity relative to established risk models
2. To determine associations between CAD severity and plaque type and:

   1. with traditional risk factors (arterial hypertension, diabetes, hypercholesterolemia, smoking)
   2. blood markers of increased cardiovascular risk
3. To determine predictive associations of between CAD with outcome (endpoint definitions in appendix)
4. To determine the risk-benefit ratio (number of subsequent interventions, complications, radiation exposure, late onset of cancer diseases, etc).

DETAILED DESCRIPTION:
Particular aims include:

1. To determine the prevalence of CAD for age, gender, ethnicity relative to established risk models
2. To determine associations between CAD severity and plaque type and:

   1. with traditional risk factors (arterial hypertension, diabetes, hypercholesterolemia, smoking)
   2. blood markers of increased cardiovascular risk
3. To determine predictive associations of between CAD with outcome (endpoint definitions in appendix)
4. To determine the risk-benefit ratio (number of subsequent interventions, complications, radiation exposure, late onset of cancer diseases, etc).

ELIGIBILITY:
Inclusion Criteria:

1. Adults (=/>18 years of age)
2. Able to provide informed consent
3. Clinical indication for cardio-CT in line with the latest clinical guidelines

Exclusion Criteria:

1. standard contraindications to CT (in line with local roles and guidelines - please see Appendix)
2. known allergy to iodinated contrast agent
3. suspected acute kidney injury
4. unstable hemodynamic status or arrhythmias
5. suspected acute coronary syndrome
6. manifest thyrotoxicosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults referred to clinical cardiac computertomography imaging
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Survival | 2 year
  number of deaths
Survival | 5 year
  number of deaths

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for experimental and translational cardiovascular imaging, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided